CLINICAL TRIAL: NCT01376167
Title: A Multi-centre, Double-blind, Randomised, Parallel-group, Active Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Tafenoquine (SB-252263, WR238605) in Subjects With Plasmodium Vivax Malaria.
Brief Title: Ph 2B/3 Tafenoquine (TFQ) Study in Prevention of Vivax Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112582; TAF112582
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-02

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine; tafenoquine; Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Tafenoquine 50mg (Experimental): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 50mg Tafenoquine will be administered on either Day 1 or Day2 depending on when eligibility is confirmed.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg; Drug: Tafenoquine 50mg
- Tafenoquine 100mg (Experimental): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 100mg Tafenoquine will be administered on either Day 1 or Day2 depending on when eligibility is confirmed.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg; Drug: Tafenoquine 100mg
- Tafenoquine 300mg (Experimental): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 300mg Tafenoquine will be administered on either Day 1 or Day2 depending on when eligibility is confirmed.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg; Drug: Tafenoquine 300mg
- Tafenoquine 600mg (Experimental): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 600mg Tafenoquine will be administered on either Day 1 or Day2 depending on when eligibility is confirmed.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg; Drug: Tafenoquine 600mg
- Primaquine 15mg (Active Comparator): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 15mg Primaquine once daily Days 2-15.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg; Drug: Primaquine 15mg
- Chloroquine only (Placebo Comparator): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered.
  Interventions: Drug: Chloroquine 600mg; Drug: Chloroquine 300mg
- Tafenoquine 300mg (Part 2) (Experimental): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 300mg Tafenoquine will be administered on either Day 1 or Day2 depending on when eligibility is confirmed.
  Interventions: Drug: Chloroquine 600mg (Part 2 ); Drug: Chloroquine 300mg (Part 2 ); Drug: Tafenoquine 300mg (Part 2)
- Primaquine 15mg (Part 2) (Active Comparator): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered. 15mg Primaquine once daily Days 2-15
  Interventions: Drug: Chloroquine 600mg (Part 2 ); Drug: Chloroquine 300mg (Part 2 ); Drug: Primaquine 15mg (Part2 )
- Chloroquine only (Part 2) (Placebo Comparator): On Day 1 and Day 2 600mg Chloroquine will be administered, on Day 3 300mg Chloroquine will be administered
  Interventions: Drug: Chloroquine 600mg (Part 2 ); Drug: Chloroquine 300mg (Part 2 )

INTERVENTIONS:
Drug: Chloroquine 600mg — 600mg Chloroquine given to each subject on Day 1 and Day2 of the trial
  Arms: Chloroquine only; Primaquine 15mg; Tafenoquine 100mg; Tafenoquine 300mg; Tafenoquine 50mg; Tafenoquine 600mg
Drug: Chloroquine 300mg — 300mg Chloroquine given to each subject on Day 3 of the trial
  Arms: Chloroquine only; Primaquine 15mg; Tafenoquine 100mg; Tafenoquine 300mg; Tafenoquine 50mg; Tafenoquine 600mg
Drug: Tafenoquine 50mg — single dose 50mg Tafenoquine given to subject on treatment arm 1 on Days 1 or 2
  Arms: Tafenoquine 50mg
Drug: Tafenoquine 100mg — single dose 100mg Tafenoquine given to subject on treatment arm 2 on Days 1 or 2
  Arms: Tafenoquine 100mg
Drug: Tafenoquine 300mg — single dose 300mg Tafenoquine given to subject on treatment arm 3 on Days 1 or 2
  Arms: Tafenoquine 300mg
Drug: Tafenoquine 600mg — single dose 600mg Tafenoquine given to subject on treatment arm 4 on Days 1 or 2
  Arms: Tafenoquine 600mg
Drug: Primaquine 15mg — 15mg Primaquine given once daily to subject on treatment arm 5 on Days 2 to 15.
  Arms: Primaquine 15mg
Drug: Chloroquine 600mg (Part 2 ) — 600mg Chloroquine given to each subject on Day 1 and Day2 of the trial.
  Arms: Chloroquine only (Part 2); Primaquine 15mg (Part 2); Tafenoquine 300mg (Part 2)
Drug: Chloroquine 300mg (Part 2 ) — 300mg Chloroquine given to each subject on Day 3 of the trial.
  Arms: Chloroquine only (Part 2); Primaquine 15mg (Part 2); Tafenoquine 300mg (Part 2)
Drug: Tafenoquine 300mg (Part 2) — single dose 300mg Tafenoquine given to subject on treatment arm 3 on Days 1 or 2.
  Arms: Tafenoquine 300mg (Part 2)
Drug: Primaquine 15mg (Part2 ) — 15mg Primaquine given once daily to subject on treatment arm 3 on Days 2 to 15.
  Arms: Primaquine 15mg (Part 2)

SUMMARY:
The purpose of this two part study is to test the safety and efficacy of Tafenoquine (with Cholorquine) as a radical cure for Plasmodium vivax (P.vivax) malaria relative to the control Chloroquine.Part 1 aims to select an efficacious and well tolerated dose that can be co-administered with Chloroquine. Part 2 will investigate the safety and efficacy of the selected dose (300 mg tafenoquine) in the treatment and radical cure of Plasmodium Vivax Malaria.

DETAILED DESCRIPTION:
Plasmodium vivax represents 50-80% of all malarial cases in Latin America and South East Asia. It is able to establish a dormant liver stage called the hypnozoite. Hypnozoite activation after initial infection can cause a relapse. Currently the only widely available drug is primaquine which requires administration over 14 days, resulting in poor compliance and treatment failure. Tafenoquine (an 8-aminoquinoline anti-malarial drug) has been shown to possess activity against all stages of the plasmodium life cycle, including the dormant stage in the liver. This is a multi-centre, double dummy, double blind, parallel group, randomized, active control study which is conducted in two parts. For both parts, subjects are treated with Chloroquine on days 1 to 3 (600mg, 600mg, and 300mg) to treat the blood stage vivax malaria. Part 1 will include at least 324 subjects and part 2 at least 600 subjects. Part 1 has 6 treatment arms, arms 1 to 4 contain different doses of Tafenoquine (50mg, 100mg, 300mg, and 600mg) dosed on day 1 or 2, arm 5 contains primaquine (15mg) dosing over 14 days (days 2-15 (15mg)) and arm 6 contains chloroquine only. The aim of this is to find a dose of Tafenoquine which meets the defined dose criteria. Based on Part 1 efficacy and safety, a single Tafenoquine dose (300 mg) will be studied in the pivotal Part 2. Part 2 contains 3 treatment arms one with the selected Tafenoquine dose (300 mg), the second arm will be 15mg Primaquine which will again be dosed over 14 days and the final arm contains chloroquine only dosed days 1-3 (600mg, 600mg, 300mg). Therefore as with Part 1, in Part 2 all subjects will receive Chloroquine. The aim of Part 2 is to investigate the safety and efficacy of the selected Tafenoquine/Chloroquine dose in the treatment and radical cure of Plasmodium vivax malaria. In addition to the Primary and Secondary endpoints stated below we will also be collecting; other efficacy endpoints (gametocyte clearance time, Recrudescence defined as any Plasmodium vivax parasitemia occurring on or before Day 29 (blood stage treatment failure), Incidence of Plasmodium falciparum malaria and Incidence of recrudescence and new Plasmodium vivax infection, determined by Polymerase Chain Reaction (PCR), safety endpoints (clinically relevant haemolysis leading to drops in haemoglobin / haematocrit or complications thereof (required transfusions, acute renal failure), changes in methaemoglobin, gastrointestinal (GI) tolerability - incidence of abdominal pain, heartburn, diarrhoea, constipation, nausea and vomiting and ophthalmic safety - incidence of corneal deposits, retinal and visual field abnormalities. Data collected at up to four centres . Additionally, the incidence and severity of adverse events and abnormal laboratory observations will be presented).Pharmacokinetic endpoints (Population pharmacokinetic parameters for tafenoquine including but not limited to oral clearance (CL/F) and volume of distribution (V/F)and Pharmacokinetic/Pharmacodynamic endpoints (e.g. tafenoquine plasma concentrations) and selected Pharmacodynamic endpoints (e.g. relapse efficacy, change in methaemoglobin) if appropriate, will be explored.

ELIGIBILITY:
Inclusion Criteria: - Positive Giemsa smear for P. vivax

* Parasite density >100 and <200,000/μL
* ≥16 years
* A female is eligible if she is non-pregnant, nonlactating and if she is of: - non-child bearing potential defined as: post-menopausal (12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone >40 mIU/mL), pre-menopausal and has had a hysterectomy or a bilateral oophorectomy (removal of the ovaries) or a bilateral tubal ligation with medical report verification, negative pregnancy test or,
* child-bearing potential, has a negative serum pregnancy test at screening, and agrees to comply with one of the following during the treatment stage of the study and for a period of 90 days after stopping study drug:
* Use of oral contraceptive, either combined or progestogen alone used in conjunction with double barrier method as defined below
* Use of an intrauterine device with a documented failure rate of <1% per year
* Use of depo provera injection (part 2)
* Double barrier method consisting of spermicide with either condom or diaphragm
* Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female.
* Complete abstinence from intercourse for 2 weeks prior to administration of study drug, throughout the study and for a period of 90 days after stopping study drug.
* A signed and dated informed consent is obtained from the subject or the subject's legal representative prior to screening.

NB Assent is obtained from subjects <18 years, where applicable and written or oral witnessed consent has been obtained from parent or guardian.

* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* Willing to be hospitalized for 3 days and return to clinic for all follow-up visits including Day 180
* QTc <450 msec at screening, based on a single QTcF value at screening (part 1 only) or as an average of triplicate Electrocardiogram obtained over a brief recording period by machine or manual over-read if first is >450 msec.- Exclusion Criteria: - Mixed malaria infections (e.g. identified by Giemsa-stained smear or rapid diagnostic test)
* Severe vivax malaria as defined by World Health Organisation criteria.
* Severe vomiting (no food or inability to take food during previous 8 hours)
* Screening haemoglobin concentration <7 g/dL.
* Glucose 6-phosphate dehydrogenase deficiency, assessed by a quantitative spectrophotometric phenotype assay:

Part 1 - Males: Any subject with an enzyme level <70% of the site median value for Glucose 6-phosphate dehydrogenase normals will be excluded. Females: Those females with a screening Hb ≥ 10 g/dL will only be excluded if their enzyme level is <70% of the site median value for Glucose 6-Phosphate dehydrogenase normals. hose females with Hb ≥7 but < 10 g/dL will be excluded if an enzyme level is not > 90% of the site median value for Glucose 6-Phosphate dehydrogenase normals.

Part 2 - Any subject with enzyme level <70% of the site median value for Glucose 6-phosphate dehydrogenase normals will be excluded

* Liver function test alanine transaminase >2x Upper Limit of Normal
* Any clinically significant concurrent illness (e.g. pneumonia, septicaemia), pre-existing conditions (e.g. renal disease, malignancy), conditions that may affect absorption of study medication (e.g. vomiting or severe diarrhea) or clinical signs and symptoms of severe cardiovascular disease (e.g. uncontrolled congestive heart failure or severe coronary artery disease). These abnormalities may be identified on the screening history and physical or laboratory examination.
* Subject has taken antimalarials (e.g. ACT, mefloquine, primaquine, chloroquine) or drugs with anti-malarial activity within the past 30 days by history.
* History of allergy to chloroquine, mefloquine, tafenoquine, primaquine or to any other 4- or 8-aminoquinolines.
* Any contraindications to chloroquine or primaquine administration including a history of porphyria, psoriasis or epilepsy (please refer to chloroquine and primaquine locally approved prescribing information).
* Subject who has previously received study medication for this protocol (all parts) or has received treatment with any other investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* History of illicit drug abuse or heavy alcohol intake within 6 months of the study.
* Subjects who have taken or will likely require the use of medications from the prohibited medication list which include the following classes: Histamine-2 blockers and antacids.
* Drugs with haemolytic potential.
* Drugs known to prolong the QTc interval

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- GSK Investigational Site, Bāndarban, Bangladesh
- Brazil (2):
  - GSK Investigational Site, Manaus, Amazonas
  - GSK Investigational Site, Porto Velho, Rondônia
- GSK Investigational Site, Oddar Meancheay Province, Cambodia
- Ethiopia (2):
  - GSK Investigational Site, Gonder
  - GSK Investigational Site, Jimma
- India (4):
  - GSK Investigational Site, Bikaner
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Secunderabad
- GSK Investigational Site, Iquitos, Loreto, Peru
- GSK Investigational Site, Rio Tuba, Bataraza, Philippines
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Tak

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lacerda MVG, Llanos-Cuentas A, Krudsood S, Lon C, Saunders DL, Mohammed R, Yilma D, Batista Pereira D, Espino FEJ, Mia RZ, Chuquiyauri R, Val F, Casapia M, Monteiro WM, Brito MAM, Costa MRF, Buathong N, Noedl H, Diro E, Getie S, Wubie KM, Abdissa A, Zeynudin A, Abebe C, Tada MS, Brand F, Beck HP, Angus B, Duparc S, Kleim JP, Kellam LM, Rousell VM, Jones SW, Hardaker E, Mohamed K, Clover DD, Fletcher K, Breton JJ, Ugwuegbulam CO, Green JA, Koh GCKW. Single-Dose Tafenoquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2019 Jan 17;380(3):215-228. doi: 10.1056/NEJMoa1710775. PMID 30650322
- [Derived] Roper DR, De la Salle B, Soni V, Fletcher K, Green JA. Abrogation of red blood cell G6PD enzyme activity through Heat treatment: development of survey material for the UK NEQAS G6PD scheme. Int J Lab Hematol. 2017 Jun;39(3):308-316. doi: 10.1111/ijlh.12627. Epub 2017 Mar 20. PMID 28318100
- [Derived] Beck HP, Wampfler R, Carter N, Koh G, Osorio L, Rueangweerayut R, Krudsood S, Lacerda MV, Llanos-Cuentas A, Duparc S, Rubio JP, Green JA. Estimation of the Antirelapse Efficacy of Tafenoquine, Using Plasmodium vivax Genotyping. J Infect Dis. 2016 Mar 1;213(5):794-9. doi: 10.1093/infdis/jiv508. Epub 2015 Oct 23. PMID 26500351
- [Derived] Tenero D, Green JA, Goyal N. Exposure-Response Analyses for Tafenoquine after Administration to Patients with Plasmodium vivax Malaria. Antimicrob Agents Chemother. 2015 Oct;59(10):6188-94. doi: 10.1128/AAC.00718-15. Epub 2015 Jul 27. PMID 26248362
- [Derived] Llanos-Cuentas A, Lacerda MV, Rueangweerayut R, Krudsood S, Gupta SK, Kochar SK, Arthur P, Chuenchom N, Mohrle JJ, Duparc S, Ugwuegbulam C, Kleim JP, Carter N, Green JA, Kellam L. Tafenoquine plus chloroquine for the treatment and relapse prevention of Plasmodium vivax malaria (DETECTIVE): a multicentre, double-blind, randomised, phase 2b dose-selection study. Lancet. 2014 Mar 22;383(9922):1049-58. doi: 10.1016/S0140-6736(13)62568-4. Epub 2013 Dec 19. PMID 24360369
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-centre, double-blind, randomized, parallel-group, active-controlled study to evaluate the efficacy, safety and tolerability of tafenoquine (TQ) in participants with Plasmodium vivax (P vivax) malaria. TAF112582 consisted of two parts-Part 1 (Phase 2 dose ranging) and Part 2 (Phase 3 pivotal). Results have been presented for Part 2.
Pre-assignment Details: A total of 683 participants were screened of which 161 failed screening and 522 participants were randomized to receive chloroquine (CQ) + 300 milligrams (mg) TQ, CQ + 15 mg primaquine (PQ) and CQ alone regimen in a ratio of 2:1:1.
Groups:
- CQ Only: Participants were administered a single oral dose of CQ 600 mg on Days 1 and 2 and CQ 300 mg on Day 3. TQ placebo was administered on Day 1 or Day 2. PQ placebo capsule was administered once daily for 14 days starting from either Day 1 or Day 2.
- TQ + CQ: Participants were administered a single oral dose of CQ 600 mg on Days 1 and Day 2 and CQ 300 mg on Day 3. Participants were dosed with TQ 300 mg either on Day 1 or Day 2. PQ placebo capsule was administered once daily for 14 days starting from either Day 1 or Day 2.
- PQ + CQ: Participants were administered a single oral dose of CQ 600 mg on Days 1 and 2 and CQ 300 mg on Day 3. Participants were dosed with TQ placebo either on Day 1 or Day 2 and PQ 15 mg was administered once daily for 14 days starting from either Day 1 or Day 2.
Period: Overall Study
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Started | 133 | 260 | 129
Completed | 129 | 250 | 123
Not Completed | 4 | 10 | 6
Not completed — Lost to Follow-up | 2 | 4 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CQ Only | TQ + CQ | PQ + CQ | Total
Number analyzed (Participants) | 133 | 260 | 129 | 522
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (14.23) | 35.0 (14.39) | 34.7 (14.26) | 35.0 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 64 | 30 | 130
  Male | 97 | 196 | 99 | 392
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American(Amer) Indian(Ind) or Alaska(Al) Native(N) | 43 | 81 | 41 | 165
  Asian-South East Asian (A) Heritage (Her) | 26 | 50 | 26 | 102
  Black or African (Afr) Amer | 14 | 28 | 13 | 55
  White-White/Caucasian(Cau)/European(Eur) Her | 3 | 4 | 2 | 9
  Multiple-Afr Amer/Afr Her/Amer Ind or Al N | 47 | 95 | 47 | 189
  Multiple-Afr Amer/Afr Her/White-White/Cau/Eur Her | 0 | 1 | 0 | 1
  Multiple-Amer Ind or Al N/A-Central/South A Her | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence-free Efficacy at 6 Months Post Dose
Description: A participant was considered to have demonstrated recurrence-free efficacy at 6 months if: a) Participant had non-zero P vivax asexual parasite count at Baseline. b) Participant showed initial clearance of P vivax parasitemia defined as two negative asexual P vivax parasite counts, with at least 6 hours between the counts, and no positive counts in the interval. c) Participant had no positive asexual P vivax parasite count at any assessment prior to or on Study Day 201 following initial parasite clearance. d) Participant did not take a concomitant medication with anti-malarial activity at any point between Study Day 1 and their last parasite assessment. e) Participant is parasite-free at 6 months. Participants were censored if they did not have P.vivax at Baseline, or took a drug with anti-malarial action despite not having malaria parasites, or did not have a 6 month assessment. The number of participants with recurrence-free efficacy at 6 months has been summarized.
Time Frame: 6 months post dose
Population: Microbiologic intent to treat (mITT) Population-all randomized participants who received at least one dose of study medication, who have at least one P vivax parasite assessment after randomization, and who have a positive parasite smear for P vivax at Baseline.
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants | 35 | 155 | 83
Statistical Analysis 1: Comparison: CQ Only vs TQ + CQ; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model — The Cox proportional hazards model was fitted with region and treatment as covariates; Hazard Ratio (HR) = 0.299, 95% CI 2-sided [0.222 to 0.404] — A hazard ratio<1 indicated a lower chance of relapse compared to CQ only
Statistical Analysis 2: Comparison: CQ Only vs PQ + CQ; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model — The Cox proportional hazards model was fitted with region and treatment as covariates; Hazard Ratio (HR) = 0.262, 95% CI 2-sided [0.178 to 0.387] — A hazard ratio<1 indicated a lower chance of relapse compared to CQ only
Statistical Analysis 3: Comparison: CQ Only vs TQ + CQ; Test type: Superiority; p < 0.001, Regression, Logistic — Logistic regression model was fitted with region and treatment as covariates. Participants with a zero P vivax asexual parasite count at Baseline were excluded from the analysis; Odds Ratio (OR) = 0.241, 95% CI 2-sided [0.152 to 0.382] — Odds ratios < 1 suggested a smaller chance of recurrence compared to CQ Only
Statistical Analysis 4: Comparison: CQ Only vs PQ + CQ; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 3]; Odds Ratio (OR) = 0.198, 95% CI 2-sided [0.117 to 0.335] — Odds ratios < 1 suggested a smaller chance of recurrence compared to CQ Only

2. Secondary Outcome: Number of Participants With Recurrence-free Efficacy at 4 Months Post Dose
Description: A participant (par) was considered to have demonstrated recurrence-free efficacy at 4 months if: a) Par had non-zero P vivax asexual parasite count at Baseline. b) Par showed initial clearance of P vivax parasitemia. c) Par had no positive asexual P vivax parasite count at any assessment prior to or on Study Day 130 following initial parasite clearance. d) Par did not take a concomitant medication with anti-malarial activity at any point between Study Day 1 and their last parasite assessment after Study Day 109 (up to and including Study Day 130). e) Par is parasite-free at 4 months defined as a negative asexual P vivax parasite count at the first parasite assessment performed after Study Day 109 (up to and including Study Day 130). Par were censored if they did not have P.vivax at Baseline, or took a drug with anti-malarial action despite not having malaria parasites or did not have a 4 month assessment. The number of par with recurrence-free efficacy at 4 months has been summarized.
Time Frame: 4 months post dose
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants | 47 | 177 | 90
Statistical Analysis 1: Comparison: CQ Only vs TQ + CQ; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model — The Cox proportional hazards model was fitted with region and treatment as covariates; Hazard Ratio (HR) = 0.271, 95% CI 2-sided [0.195 to 0.376] — A hazard ratio<1 indicated a lower chance of relapse compared to CQ only
Statistical Analysis 2: Comparison: CQ Only vs PQ + CQ; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model — The Cox proportional hazards model was fitted with region and treatment as covariates; Hazard Ratio (HR) = 0.255, 95% CI 2-sided [0.167 to 0.390] — A hazard ratio<1 indicated a lower chance of relapse compared to CQ only

3. Secondary Outcome: Time to Recurrence of P Vivax Malaria
Description: Recurrence was defined as the first confirmed presence of P vivax asexual stage parasites after clearance of initial parasitemia following CQ treatment. Time to recurrence was defined as the time (in days) from initial parasite clearance to recurrence. The time to recurrence was analyzed by the Kaplan-Meier method. NA indicates data was not available due to insufficient number of participants with events during the follow up period in the study. The median number of days to recurrence along with 95% confidence interval has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Days | 86 [63 to 109] | NA [NA to NA] — Insufficient number of participants with events during the follow up period in the study. | NA [NA to NA] — Insufficient number of participants with events during the follow up period in the study.

4. Secondary Outcome: Time to Parasite Clearance
Description: Parasite clearance time was defined as time needed to clear asexual parasite from the blood that is, parasite numbers falling below the limit of detection in the thick blood smear and remaining undetectable after 6 to 12 hours. The time taken to achieve parasite clearance was analyzed using Kaplan Meier Methodology. The median parasite clearance time along with 95% confidence interval has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Hours | 43 [41 to 48] | 45 [42 to 47] | 42 [39 to 45]

5. Secondary Outcome: Time to Fever Clearance
Description: Fever clearance time was defined as time from first dose of treatment to the time when body temperature falls to normal within Study Days 1-4 and remains normal for at least 48 hours up to the Day 8 visit. Fever clearance was considered to have been achieved once an initial temperature of more than 37.40 degree Celsius is reduced to a value less than or equal to 37.40 degree Celsius and in the absence of value more than 37.40 degree Celsius in the following 48 hours up to the Day 8 visit. The time taken to achieve fever clearance was analyzed using Kaplan Meier Methodology. The median fever clearance time along with 95% confidence interval has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Hours | 7 [5 to 14] | 7 [5 to 12] | 8 [6 to 18]

6. Secondary Outcome: Number of Participants With Hemoglobin Decline From Baseline Over First 29 Days
Description: Glucose-6-phosphate dehydrogenase deficiency (G6PD) deficiency is known to be a risk factor for hemolysis in participants treated with 8-aminoquinolines. Blood samples were collected for the evaluation of hemoglobin levels. Hemoglobin decreases of >=30% or >3 grams/deciliter (g/dL) from Baseline; or, an overall drop in hemoglobin below 6.0 g/dL in the first 15 days of the study were considered as protocol defined serious adverse events (SAEs). Number of participants with maximum hemoglobin decline from Baseline over first 29 days of study has been summarized. Safety Population consisted of all randomized participants who received at least one dose of study medication.
Time Frame: Baseline and up to Day 29
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 259 | 129
Participants
  <=20 grams/liter (g/L) | 120 | 214 | 114
  >20g/L to <=30 g/L | 11 | 31 | 12
  >30 g/L or >=30% | 2 | 14 | 3

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Potentially Related to Hemoglobin Decrease
Description: TEAEs are defined as adverse events (AEs) with an onset date and time on or after that of the start of first dose of study medication (including CQ). The number of participants with TEAEs potentially related to hemoglobin decrease has been presented.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants
  Haemoglobin decreased | 2 | 14 | 2
  Fatigue | 2 | 1 | 0
  Hyperbilirubinaemia | 1 | 0 | 0
  Pallor | 0 | 1 | 0

8. Secondary Outcome: Number of Participants Who Received Blood Transfusion
Description: The number of participants who received blood transfusion as a result of hemoglobin decline has been summarized.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Acute Renal Failure
Description: There were no participants with acute renal failure in the study.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Percent Methemoglobin
Description: Methemoglobin assessment was made with the aid of a non-invasive signal extraction pulse CO-Oximeter handheld machine (Masimo). The change from Baseline in percent methemoglobin by treatment, time and sex has been summarized. The last assessment performed prior to the first dose of study medication (CQ or randomized treatment) was considered as Baseline. Change from Baseline was calculated as the post baseline assessment minus the Baseline assessment for percent methemoglobin. Only those participants with data available at the specified data points were analyzed.
Time Frame: Baseline and up to Day 120
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent Methemoglobin
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Percent Methemoglobin
  Day 2, Male: number analyzed (Participants) | 95 | 195 | 98
  Day 2, Male | -0.18 (1.525) | -0.03 (1.246) | -0.10 (1.372)
  Day 2, Female: number analyzed (Participants) | 36 | 64 | 30
  Day 2, Female | -0.22 (0.895) | 0.10 (0.830) | -0.01 (0.438)
  Day 3, Male: number analyzed (Participants) | 97 | 195 | 99
  Day 3, Male | -0.15 (1.256) | -0.01 (1.254) | -0.02 (1.454)
  Day 3, Female: number analyzed (Participants) | 36 | 64 | 30
  Day 3, Female | -0.20 (0.902) | 0.26 (0.781) | 0.11 (0.443)
  Day 5, Male: number analyzed (Participants) | 94 | 192 | 94
  Day 5, Male | -0.28 (1.329) | 0.42 (1.633) | 1.28 (2.619)
  Day 5, Female: number analyzed (Participants) | 35 | 63 | 30
  Day 5, Female | -0.20 (0.789) | 1.37 (1.263) | 0.90 (0.885)
  Day 8, Male: number analyzed (Participants) | 97 | 191 | 96
  Day 8, Male | -0.12 (1.135) | 0.98 (1.870) | 3.01 (3.214)
  Day 8, Female: number analyzed (Participants) | 35 | 64 | 30
  Day 8, Female | -0.16 (0.857) | 2.04 (1.716) | 2.58 (2.565)
  Day 11, Male: number analyzed (Participants) | 97 | 190 | 95
  Day 11, Male | -0.07 (1.348) | 1.17 (2.074) | 3.61 (3.498)
  Day 11, Female: number analyzed (Participants) | 34 | 64 | 30
  Day 11, Female | -0.13 (0.676) | 2.13 (1.667) | 3.41 (2.659)
  Day 15, Male: number analyzed (Participants) | 96 | 189 | 94
  Day 15, Male | 0.12 (1.404) | 0.94 (1.963) | 3.51 (3.369)
  Day 15, Female: number analyzed (Participants) | 35 | 64 | 30
  Day 15, Female | -0.08 (0.684) | 1.67 (1.349) | 3.63 (2.678)
  Day 22, Male: number analyzed (Participants) | 95 | 187 | 94
  Day 22, Male | 0.07 (1.211) | 0.54 (1.431) | 1.96 (2.401)
  Day 22, Female: number analyzed (Participants) | 35 | 64 | 30
  Day 22, Female | -0.05 (0.467) | 0.93 (1.042) | 1.86 (1.494)
  Day 29, Male: number analyzed (Participants) | 95 | 190 | 93
  Day 29, Male | -0.10 (1.428) | 0.23 (1.350) | 0.58 (1.835)
  Day 29, Female: number analyzed (Participants) | 35 | 64 | 30
  Day 29, Female | -0.18 (0.927) | 0.24 (0.717) | 0.49 (0.502)
  Day 60, Male: number analyzed (Participants) | 94 | 190 | 95
  Day 60, Male | 0.44 (1.925) | -0.10 (1.362) | 0.20 (1.940)
  Day 60, Female: number analyzed (Participants) | 35 | 64 | 30
  Day 60, Female | 0.19 (1.080) | 0.03 (0.700) | 0.16 (0.620)
  Day 120, Male: number analyzed (Participants) | 93 | 187 | 93
  Day 120, Male | 0.20 (1.783) | 0.07 (1.503) | 0.37 (2.153)
  Day 120, Female: number analyzed (Participants) | 35 | 63 | 30
  Day 120, Female | 0.10 (1.332) | -0.03 (0.906) | 0.37 (1.552)

11. Secondary Outcome: Number of Participants With Gastrointestinal Disorders
Description: Gastrointestinal tolerability was analyzed by the number of par experiencing gastrointestinal disorders such as abdominal pain, heartburn, diarrhea, constipation, nausea, and vomiting. The number of participants with gastrointestinal disorders for each treatment group has been summarized.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants
  Nausea | 12 | 21 | 9
  Vomiting | 9 | 22 | 11
  Abdominal pain upper | 13 | 11 | 7
  Diarrhoea | 6 | 15 | 5
  Abdominal pain | 5 | 8 | 6
  Dyspepsia | 5 | 6 | 2

12. Secondary Outcome: Number of Participants With Keratopathy
Description: Ophthalmic assessments were carried out at pre-qualified sites (Manaus) prior to randomization and at Days 29 and 90 and at withdrawal. Assessments were carried out at Day 180 if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. The number of participants displaying keratopathy in each eye was summarized for each visit. The number of participants with new keratopathy at any time post Baseline was also reported. Ophthalmic Safety Population comprised of all participants in the Safety Population who have results from any eye assessments. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: Ophthalmic Safety Population. Day 180 was not a required follow up assessment, hence, data was not collected for most participants.
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 29 | 65 | 31
Participants
  Baseline; right eye | 0 | 0 | 0
  Baseline; left eye | 0 | 0 | 0
  Day 1; right eye | 0 | 0 | 0
  Day 1; left eye | 0 | 0 | 0
  Day 29; right eye: number analyzed (Participants) | 27 | 60 | 29
  Day 29; right eye | 0 | 0 | 0
  Day 29; left eye: number analyzed (Participants) | 27 | 60 | 29
  Day 29; left eye | 0 | 0 | 0
  Day 90; right eye: number analyzed (Participants) | 28 | 62 | 31
  Day 90; right eye | 0 | 1 | 0
  Day 90; left eye: number analyzed (Participants) | 28 | 62 | 31
  Day 90; left eye | 0 | 0 | 0
  Day 180; right eye: number analyzed (Participants) | 0 | 3 | 1
  Day 180; right eye |  | 0 | 0
  Day 180; left eye: number analyzed (Participants) | 0 | 3 | 1
  Day 180; left eye |  | 0 | 0
  Any time post Baseline; right eye | 0 | 1 | 0
  Any time post Baseline; left eye | 0 | 0 | 0

13. Secondary Outcome: Incidence of Visual Field Abnormalities Based on Best Corrected Visual Acuity Test Scores
Description: Ophthalmic assessments were carried out at pre-qualified sites (Manaus) prior to randomization and at Days 29 and 90 and at withdrawal. Assessments were carried out at Day 180 if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. Best corrected visual acuity was assessed individually for each eye. Scores were recorded as a ratio. The values were used to derive a logMAR score for statistical analysis where logMAR=-1x log10 (ratio score). The mean and standard deviation of logMAR score for each treatment group has been summarized. High scores were associated with worse vision, and low scores with better vision. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: logMAR scores
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 29 | 65 | 31
logMAR scores
  Baseline; right eye | 0.041 (0.0825) | 0.046 (0.1045) | 0.029 (0.0461)
  Baseline; left eye | 0.048 (0.0859) | 0.039 (0.0652) | 0.048 (0.1306)
  Day 29; right eye: number analyzed (Participants) | 27 | 60 | 29
  Day 29; right eye | 0.039 (0.0906) | 0.049 (0.1159) | 0.021 (0.0412)
  Day 29; left eye: number analyzed (Participants) | 27 | 60 | 29
  Day 29; left eye | 0.032 (0.0580) | 0.032 (0.0565) | 0.045 (0.1325)
  Day 90; right eye: number analyzed (Participants) | 28 | 62 | 31
  Day 90; right eye | 0.044 (0.0928) | 0.038 (0.1083) | 0.016 (0.0374)
  Day 90; left eye: number analyzed (Participants) | 28 | 62 | 31
  Day 90; left eye | 0.041 (0.0599) | 0.028 (0.0971) | 0.041 (0.1303)
  Day 180; right eye: number analyzed (Participants) | 0 | 3 | 1
  Day 180; right eye |  | 0.033 (0.0577) | 0.000 (NA) — Standard Deviation not calculable because data were only collected for 1 participant
  Day 180; left eye: number analyzed (Participants) | 0 | 3 | 1
  Day 180; left eye |  | 0.033 (0.0577) | 0.000 (NA) — Standard Deviation not calculable because data were only collected for 1 participant

14. Secondary Outcome: Number of Participants With Retinal Changes From Baseline
Description: Ophthalmic assessments were carried out at pre-qualified sites (Manaus) prior to randomization and at Days 29 and 90 and at withdrawal. Assessments were carried out at Day 180 if the Day 90 assessments showed abnormalities. The last assessment performed on the day of randomization or earlier was considered Baseline. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment. The number of participants with definite retinal change and questionable (ques) retinal change from Baseline was presented. Only those participants with data available at the specified data points were analyzed.
Time Frame: Baseline and up to Day 180
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 29 | 65 | 31
Participants
  Day 29, Definite change, right eye: number analyzed (Participants) | 24 | 53 | 23
  Day 29, Definite change, right eye | 1 | 0 | 0
  Day 29, Ques change, right eye: number analyzed (Participants) | 24 | 53 | 23
  Day 29, Ques change, right eye | 0 | 0 | 0
  Day 29, Definite change, left eye: number analyzed (Participants) | 24 | 53 | 23
  Day 29, Definite change, left eye | 1 | 0 | 0
  Day 29, Ques change, left eye: number analyzed (Participants) | 24 | 53 | 23
  Day 29, Ques change, left eye | 0 | 0 | 0
  Day 90, Definite change, right eye: number analyzed (Participants) | 24 | 48 | 23
  Day 90, Definite change, right eye | 1 | 1 | 1
  Day 90, Ques change, right eye: number analyzed (Participants) | 24 | 48 | 23
  Day 90, Ques change, right eye | 0 | 0 | 1
  Day 90, Definite change, left eye: number analyzed (Participants) | 24 | 48 | 23
  Day 90, Definite change, left eye | 1 | 1 | 0
  Day 90, Ques change, left eye: number analyzed (Participants) | 24 | 48 | 23
  Day 90, Ques change, left eye | 0 | 1 | 2
  Day 180, Definite change, right eye: number analyzed (Participants) | 1 | 7 | 0
  Day 180, Definite change, right eye | 0 | 0 |
  Day 180, Ques change, right eye: number analyzed (Participants) | 1 | 7 | 0
  Day 180, Ques change, right eye | 0 | 0 |
  Day 180, Definite change, left eye: number analyzed (Participants) | 1 | 7 | 0
  Day 180, Definite change, left eye | 0 | 0 |
  Day 180, Ques change, left eye: number analyzed (Participants) | 1 | 7 | 0
  Day 180, Ques change, left eye | 0 | 0 |

15. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant under clinical investigation, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/ birth defect, other situations and is associated with possible drug induced liver injury with hyperbilirubinemia. TEAEs is defined as AEs with an onset date and time on or after that of the start of first dose of study medication (including CQ). Number of participants with TEAEs and serious TEAEs have been presented.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants
  TEAEs | 86 | 164 | 76
  Serious TEAEs | 6 | 21 | 4

16. Secondary Outcome: Number of Participants With TEAEs by Maximum Intensity
Description: An AE is defined as any untoward medical occurrence in a participant under clinical investigation, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is defined as AEs with an onset date and time on or after that of the start of first dose of study medication (including CQ). Number of participants with AEs based on severity has been presented.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 65 | 31
Participants
  Mild or Grade 1 | 30 | 70 | 38
  Moderate or Grade 2 | 52 | 89 | 37
  Severe or Grade 3 | 3 | 2 | 1
  Grade 4 | 1 | 0 | 0
  Grade 5 | 0 | 1 | 0

17. Secondary Outcome: Number of Participants With Hematology Laboratory Data Outside the Reference Range
Description: Blood samples were collected for the evaluation of hematology parameters including eosinophils, leukocytes, lymphocytes, neutrophils, platelets, reticulocytes and methemoglobin. The number of participants with hematology laboratory data outside the extended normal range (F3) was presented. The upper and lower limits for F3 range were defined by multiplying the normal range limits by different factors. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 260 | 129
Participants
  Blood eosinophils, High: number analyzed (Participants) | 133 | 259 | 129
  Blood eosinophils, High | 18 | 38 | 28
  Blood leukocytes, Low: number analyzed (Participants) | 133 | 259 | 129
  Blood leukocytes, Low | 0 | 3 | 2
  Blood lymphocytes, Low: number analyzed (Participants) | 133 | 259 | 129
  Blood lymphocytes, Low | 7 | 4 | 0
  Blood lymphocytes, High: number analyzed (Participants) | 133 | 259 | 129
  Blood lymphocytes, High | 23 | 32 | 13
  Blood neutrophils, Low: number analyzed (Participants) | 133 | 259 | 129
  Blood neutrophils, Low | 2 | 5 | 7
  Blood platelets, Low: number analyzed (Participants) | 133 | 259 | 129
  Blood platelets, Low | 14 | 35 | 15
  Blood reticulocytes, High: number analyzed (Participants) | 133 | 259 | 129
  Blood reticulocytes, High | 72 | 141 | 85
  Methemoglobin, High | 4 | 5 | 11

18. Secondary Outcome: Number of Participants With Clinical Chemistry Laboratory Data Outside the Reference Range
Description: Blood samples were collected for the evaluation of clinical chemistry parameters including Alanine Aminotransferase (ALT), Alkaline Phosphatase (Alk. Phos), Aspartate Aminotransferase (AST), bilirubin, creatine kinase, creatinine, glomerular filtration rate (GFR), indirect bilirubin and urea. The number of participants with clinical chemistry laboratory data outside the extended normal range (F3) was presented. The upper and lower limits for F3 range were defined by multiplying the normal range limits by different factors. High and low indicated that the participants had values flagged as high and low respectively for the particular parameter any time on-treatment. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
Number analyzed (Participants) | 133 | 259 | 129
Participants
  ALT, High | 11 | 10 | 5
  Alk Phos, High | 3 | 1 | 1
  AST, High | 5 | 7 | 2
  Bilirubin, High | 18 | 23 | 12
  Creatine kinase, High | 8 | 5 | 8
  Creatinine, High | 0 | 1 | 0
  GFR, Low | 0 | 1 | 0
  Indirect bilirubin | 11 | 22 | 8
  Urea, High | 42 | 85 | 46

19. Secondary Outcome: Cost Associated With Recurrence Episode of P Vivax Malaria
Description: Health outcomes were evaluated based on the total costs spent on treatment, transport, medication and tests. The cost was summarized according to the place at which the participant went to for care (drug shop, trial clinic, other clinic, hospital (inpatient/outpatient), traditional healer, other). The reported costs by type and by site has been summarized. Where costs have not been reported at a visit, the number of participants analyzed is given as 0. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: US Dollars (USD)
Groups:
- First Malaria Recurrence: Participants from all treatment arms (CQ only, CQ+TQ and PQ+TQ) with a recurrence episode of malaria were included.
- First Malaria Recurrence Follow-up: Participants from all treatment arms (CQ only, CQ+TQ and PQ+TQ) who had a follow-up visit for recurrence episode of malaria were included.
Arm/Group | First Malaria Recurrence | First Malaria Recurrence Follow-up
Number analyzed (Participants) | 193 | 193
US Dollars (USD)
  Brazil (Drug shop for care): number analyzed (Participants) | 2 | 0
  Brazil (Drug shop for care) | 4.76 (3.24) |
  Brazil (Enrollment clinic for care): number analyzed (Participants) | 59 | 72
  Brazil (Enrollment clinic for care) | 6.17 (2.39) | 6.15 (2.14)
  Brazil (other location for care): number analyzed (Participants) | 1 | 0
  Brazil (other location for care) | 4.23 (0) |
  Peru (Drug shop for care): number analyzed (Participants) | 8 | 0
  Peru (Drug shop for care) | 1.47 (1.30) |
  Peru (Enrollment clinic for care): number analyzed (Participants) | 61 | 63
  Peru (Enrollment clinic for care) | 8.78 (7.94) | 8.54 (8.52)
  Peru (Attended another clinic): number analyzed (Participants) | 7 | 44
  Peru (Attended another clinic) | 2.71 (4.69) | 3.94 (1.42)
  Peru (Other location for care): number analyzed (Participants) | 15 | 1
  Peru (Other location for care) | 0.72 (0.41) | 1.30 (0)
  Thailand (Drug shop for care): number analyzed (Participants) | 1 | 0
  Thailand (Drug shop for care) | 4.60 (0) |
  Thailand (Enrollment clinic for care): number analyzed (Participants) | 13 | 0
  Thailand (Enrollment clinic for care) | 19.15 (10.60) |
  Thailand (In-hospital care): number analyzed (Participants) | 1 | 0
  Thailand (In-hospital care) | 6.13 (0) |

20. Secondary Outcome: Cost Incurred With Purchase of Medications Associated With Recurrence Episode of Malaria
Description: Health outcomes were evaluated based on the cost of medications purchased. The reported total medication cost for paracetamol associated with recurrence episode of P vivax malaria has been reported by site. Where costs have not been reported at a visit, the number of participants analyzed is given as 0. Medications recorded as "Other" and medications without costs are excluded from the analysis. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | First Malaria Recurrence | First Malaria Recurrence Follow-up
Number analyzed (Participants) | 29 | 3
USD
  Peru, n=23, 3: number analyzed (Participants) | 23 | 3
  Peru, n=23, 3 | 0.49 (0.1941) | 0.32 (1)
  Brazil, n=6, 0: number analyzed (Participants) | 6 | 0
  Brazil, n=6, 0 | 1.70 (0.144) |

21. Secondary Outcome: Time Lost by Participants or Care Givers From Normal Occupation
Description: Health outcomes were evaluated based on total time lost by participants or care givers due to an episode of malaria. The reported time lost due to recurrence episode of P vivax malaria has been summarized by category and by site. Where categories by site have not been reported at a visit, the number of participants analyzed is given as 0. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Days
Arm/Group | First Malaria Recurrence | First Malaria Recurrence Follow-up
Number analyzed (Participants) | 193 | 188
Days
  Brazil, Housework: number analyzed (Participants) | 16 | 15
  Brazil, Housework | 1 | 0
  Brazil, Farming: number analyzed (Participants) | 5 | 4
  Brazil, Farming | 8 | 0
  Brazil, paid employment: number analyzed (Participants) | 44 | 43
  Brazil, paid employment | 8 | 0
  Brazil, Other: number analyzed (Participants) | 17 | 16
  Brazil, Other | 3 | 5
  Cambodia, Farming: number analyzed (Participants) | 12 | 12
  Cambodia, Farming | 17 | 24
  Ethiopia, Housework: number analyzed (Participants) | 3 | 3
  Ethiopia, Housework | 4 | 3
  Ethiopia, Farming: number analyzed (Participants) | 2 | 2
  Ethiopia, Farming | 2.5 | 3
  Ethiopia, Student: number analyzed (Participants) | 2 | 2
  Ethiopia, Student | 3 | 0
  Ethiopia, Paid employment: number analyzed (Participants) | 4 | 4
  Ethiopia, Paid employment | 2 | 4
  Ethiopia, Other: number analyzed (Participants) | 3 | 3
  Ethiopia, Other | 1 | 7
  Peru, Housework: number analyzed (Participants) | 21 | 21
  Peru, Housework | 24 | 29
  Peru, Farming: number analyzed (Participants) | 14 | 14
  Peru, Farming | 19 | 28
  Peru, Student: number analyzed (Participants) | 2 | 2
  Peru, Student | 1 | 6
  Peru, Paid employment: number analyzed (Participants) | 6 | 6
  Peru, Paid employment | 6 | 8.5
  Peru, Other: number analyzed (Participants) | 20 | 20
  Peru, Other | 26 | 32
  Philippines, Farming: number analyzed (Participants) | 1 | 0
  Philippines, Farming | 0 |
  Thailand, paid employment: number analyzed (Participants) | 14 | 14
  Thailand, paid employment | 20 | 0
  Thailand, Other: number analyzed (Participants) | 2 | 2
  Thailand, Other | 1 | 0

22. Secondary Outcome: Number of Participants With Action Taken to Treat Recurrence Episode of P Vivax Malaria
Description: Health outcomes were evaluated based on the actions taken by the participants to treat recurrence episode of P vivax malaria. The reported action taken by site is summarized. Where no action by site have been reported at a visit, the number of participants analyzed is given as 0. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to Day 180
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | First Malaria Recurrence | First Malaria Recurrence Follow-up
Number analyzed (Participants) | 193 | 188
Participants
  Brazil, Nothing: number analyzed (Participants) | 86 | 81
  Brazil, Nothing | 21 | 5
  Brazil, Drug shop: number analyzed (Participants) | 86 | 81
  Brazil, Drug shop | 2 | 0
  Brazil, Trial clinic: number analyzed (Participants) | 86 | 81
  Brazil, Trial clinic | 62 | 76
  Brazil, Other: number analyzed (Participants) | 86 | 81
  Brazil, Other | 2 | 0
  Cambodia, Nothing: number analyzed (Participants) | 13 | 14
  Cambodia, Nothing | 13 | 14
  Ethiopia, Nothing: number analyzed (Participants) | 14 | 14
  Ethiopia, Nothing | 12 | 13
  Ethiopia, Another clinic: number analyzed (Participants) | 14 | 14
  Ethiopia, Another clinic | 1 | 0
  Ethiopia, Other: number analyzed (Participants) | 14 | 14
  Ethiopia, Other | 1 | 0
  Ethiopia, Trial clinic: number analyzed (Participants) | 14 | 14
  Ethiopia, Trial clinic | 0 | 1
  Peru, Nothing: number analyzed (Participants) | 63 | 63
  Peru, Nothing | 1 | 0
  Peru, Drug shop: number analyzed (Participants) | 63 | 63
  Peru, Drug shop | 8 | 0
  Peru, Trial clinic: number analyzed (Participants) | 63 | 63
  Peru, Trial clinic | 61 | 63
  Peru, Another clinic: number analyzed (Participants) | 63 | 63
  Peru, Another clinic | 10 | 54
  Peru, Other: number analyzed (Participants) | 63 | 63
  Peru, Other | 15 | 1
  Philippines, Nothing: number analyzed (Participants) | 1 | 0
  Philippines, Nothing | 1 |
  Thailand, Nothing: number analyzed (Participants) | 16 | 16
  Thailand, Nothing | 1 | 16
  Thailand, Drug shop: number analyzed (Participants) | 16 | 16
  Thailand, Drug shop | 1 | 0
  Thailand, Trial clinic: number analyzed (Participants) | 16 | 16
  Thailand, Trial clinic | 13 | 0
  Thailand, In hospital: number analyzed (Participants) | 16 | 16
  Thailand, In hospital | 1 | 0

23. Secondary Outcome: Oral Clearance (CL/F) of TQ
Description: Apparent population oral clearance of TQ
Time Frame: Day 2, Day 8, Day 15, Day 29 and Day 60
Population: Safety Population
Measure: Median (90% Confidence Interval); unit: Liters per hour
Groups:
- Participants in TQ Only Arms: TQ only arms
Arm/Group | Participants in TQ Only Arms
Number analyzed (Participants) | 259
Liters per hour | 2.96 [2.87 to 3.05]

24. Secondary Outcome: Volume of Distribution (Vc/F) of TQ
Description: Apparent population central volume of distribution of TQ
Time Frame: Day 2, Day 8, Day 15, Day 29 and Day 60
Population: Safety Population
Measure: Median (90% Confidence Interval); unit: Liters
Arm/Group | Participants in TQ Only Arms
Number analyzed (Participants) | 259
Liters | 915 [879 to 956]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the follow up contact (Up to Day 180)
Description: Safety Population comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | CQ Only | TQ + CQ | PQ + CQ
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/260 | 0/129
Serious Adverse Events (participants affected / at risk) | 6/133 | 21/260 | 4/129
Other Adverse Events (participants affected / at risk) | 72/133 | 119/260 | 56/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CQ Only (N=133) | TQ + CQ (N=260) | PQ + CQ (N=129)
Haemoglobin decreased (Investigations) | 2 (2) | 14 (14) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CQ Only (N=133) | TQ + CQ (N=260) | PQ + CQ (N=129)
Nausea (Gastrointestinal disorders) | 12 (13) | 21 (22) | 8 (8)
Vomiting (Gastrointestinal disorders) | 9 (10) | 22 (22) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 13 (13) | 11 (14) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 14 (14) | 4 (4)
Headache (Nervous system disorders) | 19 (23) | 27 (34) | 10 (13)
Dizziness (Nervous system disorders) | 11 (13) | 25 (30) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (23) | 34 (35) | 14 (14)
Nasopharyngitis (Infections and infestations) | 7 (7) | 19 (19) | 9 (11)
Pharyngitis (Infections and infestations) | 4 (4) | 13 (14) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (24) | 15 (15) | 10 (11)
Blood creatine phosphokinase increased (Investigations) | 8 (9) | 10 (10) | 7 (7)
Alanine aminotransferase increased (Investigations) | 8 (8) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.